CLINICAL TRIAL: NCT04777214
Title: A Blinded Randomized Sham-Controlled Incomplete Crossover Trial of Low-Frequency Contralesional Repetitive Transcranial Magnetic Stimulation in the Treatment of Aphasia in Patients With Chronic Stroke
Brief Title: TMS in Aphasia Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, H. Branch Coslett, Professor of Neurology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 805362
Record Dates: First submitted 2021-02-02; First posted 2021-03-02 (Actual); Results first posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-04

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: The study involves two arms. The study involves a sham treatment control for half of the patients; all patients randomized to the sham treatment will be enrolled in the treatment phase after completing the sham treatment. Patients will be randomly assigned to the treatment arm or the sham treatment arm of the study. There are 3 phases: a pre-treatment evaluation phase in which baseline language and imaging data are obtained and the optimal site for stimulation is determined; a treatment phase during which TMS is delivered on 10 occasions; and a post-treatment phase during which effects of the treatment will be assessed using behavioral measures as well as fMRI at 2 and 6-months. Participants in the sham arm will undergo the same behavioral testing, MRI, and fMRI that will be administered in the treatment protocol. After the 2-month follow up visit, patients in the sham arm will be told that they did not receive real TMS and will be offered the opportunity to enter the treatment arm.
Who Masked: Participant, Care Provider
Masking Description: The procedure for localizing the site of stimulation and TMS administration will be identical to the treatment arm, except the coil will be rotated 90 degrees during the process/administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active TMS (Active Comparator): There are 10 TMS sessions over 2 consecutive weeks in which 20 minutes (1200 pulses) of 1 Hz active TMS are delivered to a previously determined optimal response site in right frontal lobe.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham TMS (Sham Comparator): There are 10 TMS sessions over 2 consecutive weeks in which 20 minutes (1200 pulses) of 1 Hz TMS are delivered, however, the coil will be rotated 90 degrees during stimulation.
  Interventions: Device: Sham TMS

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Active TMS will be at 90% motor threshold
  Arms: Active TMS
Device: Sham TMS — Sham TMS will be administered
  Arms: Sham TMS

SUMMARY:
Stroke often causes substantial problems in speaking or understanding speech. Treatments for these problems are currently very limited. Limited studies to date suggest that repetitive Transcranial Magnetic Stimulation (TMS) to the side of the brain opposite to the side on which the stroke occurred may improve language function. The investigators are testing this hypothesis by giving daily 20 minute sessions of repeated TMS to the right (unaffected) side of the brain; the investigators test language function with a variety of tests both before and after the treatment with TMS and subjects are required to undergo functional MRI scans before and after treatment. TMS is a procedure in which a coil is placed next to the head of the subject and an electrical current passes through the coil causing a magnetic field that, in turn, causes a small electric current in the portion of the brain underneath the coil.

ELIGIBILITY:
Inclusion Criteria:

* Aphasic patients will have had single, unilateral left hemisphere ischemic stroke, which spared the supplementary motor area (SMA)
* With the exception of lacunar infarcts less than ≤ 1.5 cm (as measured by neuroimaging), the stroke causing the patients' impairments must be the only stroke.
* Aphasic patients will be at least 6 months post-stroke and have mild-severe, non-fluent speech
* Participants must be able to understand the nature of the study, and give informed consent

Exclusion Criteria:

* Patients with more than one stroke
* Primary hemorrhagic stroke. Note: It is recognized that some ischemic strokes may have a minor amount of hemosiderin in the parenchyma. If this occurs, this is not considered a "hemorrhagic stroke" referred to in this exclusion criterion.
* Intracranial metallic bodies from prior neurosurgical procedure
* Signs of increased intracranial pressure as assessed by ophthalmic exam and patient symptoms
* Implanted pacemaker, medication pump, vagal nerve stimulator, deep brain stimulator, TENS unit or ventriculoperitoneal shunt
* History of seizure or unexplained loss of consciousness during the year prior to the initiation of the study
* Pregnancy. If the patient cannot rule out pregnancy then a pregnancy test will be conducted prior to inclusion into the study
* Family history of epilepsy
* Acute, unstable medical conditions
* History of substance abuse within the last 6 months
* Abnormal neurologic exam other than as signs of the condition studied in the present protocol
* History of known structural brain abnormality other than as signs of the condition studied in the present protocol
* History of tinnitus
* History of bipolar disorder
* Consumption of medicines known to lower the seizure threshold
* History of head injury with unconsciousness lasting more than 5 minutes
* Previous brain surgery
* Other medical or neurologic conditions, aside from stroke, in which the likelihood of developing a seizure is known to be increased
* Other medical or neurologic conditions, in which a seizure would be particularly harmful
* Significant cardiac disease
* Intracardiac lines of any type
* Current serious or unstable medical illness, including renal, hepatic, cardiovascular, gastrointestinal, endocrinologic, neurologic, immunologic, or hematological disease, that could require admission to a hospital within 3 months, or that death is anticipated within 3 years, or that requires daily supervision by a health professional
* Administration of any investigational drug within 5 half-lives of the drug prior to testing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-06-26 (Actual); Primary Completion 2011-08-30 (Actual); Study Completion 2011-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Branch Coslett, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were assessed against the study inclusion and exclusion criteria. Eligible patients then underwent language tests before and after 6 ten minute sessions of rTMS to determine if there was a right hemisphere cortical region which, when suppressed with 1 Hz rTMS, resulted in significantly improved naming. If no benefit was observed from stimulation, the patient did not continue on to the treatment phase.
Groups:
- Sham TMS: There are 10 TMS sessions over 2 consecutive weeks in which 20 minutes (1200 pulses) of 1 Hz TMS are delivered, however, the coil will be rotated 90 degrees during stimulation.
  Sham TMS: Sham TMS will be administered
  at least 2 months later, patients then receive Active TMS if they so choose. There are 10 TMS sessions over 2 consecutive weeks in which 20 minutes (1200 pulses) of 1 Hz active TMS are delivered to a previously determined optimal response site in right frontal lobe.
  Repetitive Transcranial Magnetic Stimulation: Active TMS will be at 90% motor threshold
Period: Initial Randomization
Arm/Group | Active TMS | Sham TMS
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Sham Crossover to Active TMS Arm
Arm/Group | Active TMS | Sham TMS
Started (Only patients initially randomized to Sham arm continue on the crossover arm. Patients initially randomized to Active arm do not crossover to Sham arm) | 0 | 5
Completed | 0 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active TMS | Sham TMS | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (7.09) | 62.6 (10.14) | 61.6 (8.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Boston Naming Test
Description: The Boston Naming Test is an assessment of confrontation naming, where a score ranges from 0 (no items named correctly) to 36 (all items named correctly)
Time Frame: Baseline, 2 months and 6-months after the last rTMS treatment session
Population: 9 participants completed the Active TMS arm and were available for follow-up at 2- and 6- months post treatment.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Groups:
- Active TMS 2-month Follow-Up: There are 10 TMS sessions over 2 consecutive weeks in which 20 minutes (1200 pulses) of 1 Hz active TMS are delivered to a previously determined optimal response site in right frontal lobe.
  Repetitive Transcranial Magnetic Stimulation: Active TMS will be at 90% motor threshold
  Outcome measures are then assessed 2 months after TMS treatment sessions.
- Active TMS 6-month Follow-Up: There are 10 TMS sessions over 2 consecutive weeks in which 20 minutes (1200 pulses) of 1 Hz active TMS are delivered to a previously determined optimal response site in right frontal lobe.
  Repetitive Transcranial Magnetic Stimulation: Active TMS will be at 90% motor threshold
  Outcome measures are then assessed 6 months after TMS treatment sessions.
Arm/Group | Active TMS 2-month Follow-Up | Active TMS 6-month Follow-Up
Number analyzed (Participants) | 9 | 9
percent change from baseline | 10.3 (20.0) | 37.7 (31.2)

2. Other Pre Specified Outcome: Picture Description of the Boston Diagnostic Aphasia Exam
Description: The picture description of the Boston Diagnostic Aphasia Exam is a measurement of spontaneous speech, elicited by a picture description. It is not a scale. Quantitative Production Analysis (QPA) is used to analyze the production of words related to the picture stimulus. Total number of Narrative Words produced, defined as total words minus stereotyped utterances, task-related comments, or comments cued by administrator, was determined using QPA as a measure of discourse productivity.
Time Frame: Baseline and 2 months after the last rTMS treatment session
Population: Comparison of total narrative word output change between baseline and 2-months between Active arm and Sham Arm. Active TMS arm includes both 5 participants initially randomized to Active TMS arm, plus 5 people who crossed over to Active arm after Sham arm.
Measure: Mean (Standard Deviation); unit: change in number of words from baseline
Arm/Group | Active TMS | Sham TMS
Number analyzed (Participants) | 10 | 5
change in number of words from baseline | 10.4 (16.3) | 1.2 (15.0)

3. Other Pre Specified Outcome: Boston Diagnostic Aphasia Exam - Word Discrimination Subtest
Description: The Boston Diagnostic Aphasia Exam - Word Discrimination Subtest is an assessment of auditory comprehension via word discrimination, where a score ranges from 0 (no items correct) to 72 (all items correct)
Time Frame: Baseline and 2 months after the last rTMS treatment session
Population: Comparison of percent change in outcome between baseline and 2-months between Active arm and Sham Arm. Active TMS arm includes both 5 participants initially randomized to Active TMS arm, plus 5 people who crossed over to Active arm after Sham arm.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Active TMS | Sham TMS
Number analyzed (Participants) | 10 | 5
Percent change from baseline | 1.78 (6.83) | 0.32 (1.51)

4. Other Pre Specified Outcome: Boston Diagnostic Aphasia Examination - Commands Subtest
Description: The Boston Diagnostic Aphasia Examination - Commands Subtest is an assessment of auditory comprehension via command following, where a score ranges from 0 (no items correctly performed) to 15 (all items correctly performed). Percent change was calculated by taking the mean performance at 2-months after rTMS treatment and subtracting mean performance at baseline, then dividing by the mean baseline performance and multiplying by 100.
Time Frame: Baseline and 2 months after the last rTMS treatment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Active TMS | Sham TMS
Number analyzed (Participants) | 10 | 5
percent change from baseline | 2.22 (12.08) | 8.00 (10.26)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from enrollment in the study to 30 days following administration of rTMS treatment, on average 303.3 days.
Description: An adverse event is any symptom, sign, illness or experience that develops or worsens in severity during the course of the study. A serious adverse event is any AE that is: fatal, life-threatening, requires or prolongs hospital stay, results in persistent or significant disability or incapacity, a congenital anomaly or birth defect, an important medical event Important medical events are those that may not be immediately life threatening, but are clearly of major clinical significance.
Arm/Group | Active TMS | Sham TMS
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No